CLINICAL TRIAL: NCT03583515
Title: Self-Determination Theory as A Framework For Evaluating Within-Person Effects Of Personalized Normative Feedback On Drinking
Brief Title: Evaluating Within-Person and Between-Person Effects Of A Personalized Normative Feedback Intervention On Drinking As They Are Moderated By Self-Determination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, C. Raymond Knee, Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1F31AA026195-01A1 (NIH); 1F31AA026195-01A1 (NIH)
Record Dates: First submitted 2018-06-01; First posted 2018-07-11 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Half of participants will be randomly assigned to receive personalized normative feedback about their drinking. The other half will be randomly assigned to receive control feedback about social media use.
Who Masked: Participant, Investigator
Masking Description: Participants will be assigned to and receive feedback via the computer. Once they have received feedback a research assistant will print this feedback for them to take home. At this time, research assistants will become unblinded to condition, but will not administer any new procedures other than answering participant questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol-Specific Personalized Normative Feedback (Experimental): Participants will receive feedback about their average number of days on which alcohol was consumed, average drinks per occasion, and average number of drinks per week. This feedback will include the participant's averages reported at baseline, the participant's descriptive norm of others' averages (what they think others drank), and actual others' drinking. Feedback will be about other students at their university of the same sex.
  Interventions: Behavioral: Alcohol-Specific Personalized Normative Feedback
- Social Media Personalized Normative Feedback (Placebo Comparator): Participants will receive feedback about their number of hours texting, on social media websites, and playing video games. This feedback will include the participant's averages reported at baseline, the participant's descriptive norm of others' averages (what they think others did), and actual others' behavior. Feedback will be about other students at their university of the same sex.
  Interventions: Behavioral: Social Media Personalized Normative Feedback

INTERVENTIONS:
Behavioral: Alcohol-Specific Personalized Normative Feedback — Participants will receive personalized normative feedback about drinking.
  Arms: Alcohol-Specific Personalized Normative Feedback
Behavioral: Social Media Personalized Normative Feedback — Participants will receive personalized normative feedback about social media use.
  Arms: Social Media Personalized Normative Feedback

SUMMARY:
This study evaluates within-person and between-person effects of a personalized normative feedback intervention and injunctive norms as they are altered by self-determination in heavy drinkers. Half of participants will receive personalized normative feedback and the other half will receive control feedback about media use habits.

ELIGIBILITY:
Inclusion Criteria:

* Student at the University of Houston
* Above 18 years of age
* Heavy drinker (more than 4 drinks [women] or 5 drinks [men] on a single occasion in the last 2.5 weeks and drinks, on average, at least once per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Between-Person Self-Determination by PNF Interaction Predicting Consumption | 2-4 Weeks
  A structural equation model will be fit with baseline consumption, self-determination, intervention condition, and the interaction between self-determination and condition predicting follow-up alcohol consumption. Consumption will be measured with the Alcohol Consumption Index, Quantity-Frequency-Peak Alcohol Use Index, and the Daily Drinking Questionnaire. These scales will be used as indicators of a single latent consumption variable. That latent consumption measure will be the outcome of interest.
Within-Person Self-Determination by PNF Interaction Predicting Consumption | 17 Days
  A multilevel model will be fit with baseline consumption, daily self determination, intervention condition, and the interaction between condition and daily self-determination predicting daily alcohol consumption. Consumption will be measured as the number of drinks consumed the previous evening.

SECONDARY OUTCOMES:
Between-Person Self-Determination by PNF Interaction Predicting Alcohol-Related Problems | 2-4 Weeks
  A structural equation model will be fit with baseline consumption, alcohol-related problems, self-determination, intervention condition, and the interaction between self-determination and condition predicting follow-up alcohol-related problems. Alcohol-related problems will be measured with the Rutgers Alcohol Problems Index and the Young Adult Alcohol Consequences Questionnaire. Each of these problems measures will be split to form two indicators (for a total of four problems indicators) for an overall problems latent variable. This problems latent variable will then be used as the outcome of interest.
Within-Person Self-Determination by PNF Interaction Predicting Alcohol-Related Problems | 17 Days
  A multilevel model will be fit with baseline consumption, daily self determination, intervention condition, and the interaction between condition and daily self-determination predicting daily alcohol alcohol-related problems. Alcohol-related problems will be measured with a checklist of non-overlapping items from the Rutgers Alcohol Problems Index and the Young Adult Alcohol Consequences Questionnaire. This combined checklist will be used to create the overall problems outcome of interest.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Informed Consent Form Analytic Code De-Identified Data
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available within a year of study completion.
Access Criteria: Data will be available upon request.